CLINICAL TRIAL: NCT02606500
Title: Efficacy of Corifollitropin Alfa in Obese Women in Terms of Clinical and Molecular Parameters of IVF Success
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tanja Burnik Papler, Principal investigator Tanja Burnik Papler, MD; PhD, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck-01
Record Dates: First submitted 2015-11-06; First posted 2015-11-17 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elonva 150 mcg (Experimental): Elonva 150 mcg intramuscular daily obese
  Interventions: Drug: Elonva
- Elonva 100 mcg (Active Comparator): Elonva 100 mcg intramuscular daily normal weight
  Interventions: Drug: Elonva

INTERVENTIONS:
Drug: Elonva — 20 obese women will be the study group and 20 normal weighing women will be the control group. Both groups will receive 150 mcg of Elonva for controlled ovarian hyperstimulation (COH). Gonadotropin-releasing hormone (GnRH) antagonist will be used to prevent premature luteinizing hormone (LH) surge. Additional daily doses of 200 IU of recombinant follicle stimulating hormone (rFSH) will be used if necessary. Human chorionic gonadotropin (hCG) will be used for oocyte maturation. 2 mature follicles will be aspirated separately in each patient. Cumulus cell (CC) samples will be collected and stored on -80 oC for subsequent analysis. Clinical and molecular parameters of IVF success will be assessed and compared between the groups.
  The exclusion criteria will be: polycystic ovary syndrome, severely abnormal sperm parameters, and age > 38 years.

SUMMARY:
The aim of the present study is to determine, whether clinical efficacy of 150 mcg of Corifollitropin alfa is the same in normal weighing and obese women. Furthermore, investigators want to determine whether oocytes retrieved from normal weighing and obese women, after COH using 150 mcg of Corifollitropin alfa, are of same quality on the molecular level.

DETAILED DESCRIPTION:
The dosage of Corifollitropin alfa used for controlled ovarian hyperstimulation (COH) is adjusted according to the patient's body weight. Meaning, in women with a body weight ≤ 60 kg, a single dose of 100 mcg of Corifollitropin alfa is administered for COH and in women with a body weight > 60 kg, a single dose of 150 micrograms of Corifollitropin alfa is administered for COH. These two protocols are comparable in safety and efficacy of follicular stimulation.

On the other hand, knowledge about the clinical efficacy of 150 mcg of Corifollitropin alfa in obese women (BMI>30 kg/m2) is lacking.

Cumulus cells (CC) surround the oocyte and bi-directional communication between oocyte and CC is necessary for the development of mature and quality oocytes. It has been proposed, that analysis of genes, expressed in CC, can serve as an objective indicator of the oocyte's maturity and developmental potential. Expression of genes in CC as hyaluronan synthase 2 (HAS2), follicle-stimulating hormone receptor (FSHR), versican (VCAN), progesterone receptor (PR), vascular endothelial growth factor C (VEGFC), serine protease inhibitor E2 (SERPINE2), glutathione peroxidase (GPX3), pentraxin 3(PTX3) was reported to correlate with oocyte maturity and developmental potential.

The effect of Corifollitropin alfa on expression of these genes however, is unknown.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2
* BMI 18.5-24.9 kg/m2

Exclusion Criteria:

* polycystic ovary syndrome, severely abnormal sperm parameters, and age > 38 years

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eda Vrtacnik Bokal, professor, Study Chair — Head of the department of Human reproduction
Locations (1):
- Division of gynecology, Department of human reproduction, Ljubljana, Slovenia

REFERENCES:
- [Background] Burnik Papler T, Vrtacnik Bokal E, Maver A, Kopitar AN, Lovrecic L. Transcriptomic Analysis and Meta-Analysis of Human Granulosa and Cumulus Cells. PLoS One. 2015 Aug 27;10(8):e0136473. doi: 10.1371/journal.pone.0136473. eCollection 2015. PMID 26313571
- [Background] Burnik Papler T, Vrtacnik Bokal E, Maver A, Lovrecic L. Specific gene expression differences in cumulus cells as potential biomarkers of pregnancy. Reprod Biomed Online. 2015 Apr;30(4):426-33. doi: 10.1016/j.rbmo.2014.12.011. Epub 2015 Jan 12. PMID 25682305
- [Background] Burnik Papler T, Vrtacnik Bokal E, Lovrecic L, Kopitar AN, Maver A. No specific gene expression signature in human granulosa and cumulus cells for prediction of oocyte fertilisation and embryo implantation. PLoS One. 2015 Mar 13;10(3):e0115865. doi: 10.1371/journal.pone.0115865. eCollection 2015. PMID 25769026
- [Background] Devjak R, Fon Tacer K, Juvan P, Virant Klun I, Rozman D, Vrtacnik Bokal E. Cumulus cells gene expression profiling in terms of oocyte maturity in controlled ovarian hyperstimulation using GnRH agonist or GnRH antagonist. PLoS One. 2012;7(10):e47106. doi: 10.1371/journal.pone.0047106. Epub 2012 Oct 17. PMID 23082142
- [Background] Vrtacnik-Bokal E, Virant Klun I, Verdenik I. Follicular oestradiol and VEGF after GnRH antagonists or GnRH agonists in women with PCOS. Reprod Biomed Online. 2009 Jan;18(1):21-8. doi: 10.1016/s1472-6483(10)60420-8. PMID 19146765

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: 35 obese women (BMI ≥ 30 kg/m2) were included to the study group. 150 mcg of Elonva for controlled ovarian hyperstimulation (COH) on day 2 or 3 of menstrual cycle. GnRH antagonist was used to prevent premature LH surge. Additional daily doses of 200 IU of rFSH were used if necessary to achieve optimal ovarian stimulation. hCG was used to induce final oocyte maturation. Follicles were aspirated separately in each patient. Cumulus cells (CC) samples of the first 2 aspirated follicles were collected and stored on -80 oC for subsequent analyses. Clinical IVF parameters were assessed and compared between the groups. Also, gene expression analyses of CC were performed using quantitative real-time PCR.
  Inclusion criteria for the study group were: first or second IVF cycle, BMI ≥ 30 kg/m2, tubal factor of infertility, normal partner's spermiogram.
- Control Group: 35 normal weighing women (BMI 19 - 24.9 kg/m2) were included to the study group. 150 mcg of Elonva for controlled ovarian hyperstimulation (COH) on day 2 or 3 of menstrual cycle. GnRH antagonist was used to prevent premature LH surge. Additional daily doses of 200 IU of rFSH were used if necessary to achieve optimal ovarian stimulation. hCG was used to induce final oocyte maturation. Follicles were aspirated separately in each patient. Cumulus cells (CC) samples of the first 2 aspirated follicles were collected and stored on -80 oC for subsequent analyses. Clinical IVF parameters were assessed and compared between the groups. Also, gene expression analyses of CC were performed using quantitative real-time PCR.
  Inclusion criteria for the control group were: first or second IVF cycle, normal BMI (19 - 24.9 kg/m2), tubal factor of infertility and normal partner's spermiogram.
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: 35 normal weighing women (BMI 19 - 24.9 kg/m2) were included to the study group. 150 mcg of Elonva for controlled ovarian hyperstimulation (COH) on day 2 or 3 of menstrual cycle. GnRH antagonist was used to prevent premature LH surge. Additional daily doses of 200 IU of rFSH were used if necessary to achieve optimal ovarian stimulation. hCG was used to induce final oocyte maturation. Follicles were aspirated separately in each patient. Cumulus cells (CC) samples of the first 2 aspirated follicles were collected and stored on -80 oC for subsequent analyses. Clinical IVF parameters were assessed and compared between the groups. Also, gene expression analyses of CC were performed using quantitative real-time PCR.
  Inclusion criteria for the control group were: first or second IVF cycle, normal BMI (19 - 24.9 kg/m2), tubal factor of infertility and normal partner's spermiogram.
  s.
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 30.3 (3.9) | 31.5 (3.6) | 30.9 (3.7)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Only women were included in the study.
  Participants
    Women | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 35 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Slovenia | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved Per Patient
Description: Number of oocytes obtained in the study group was compared to the number of oocytes obtained in the control group
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 35 | 35
Oocytes | 11.3 (7.5) | 12.4 (7.4)
Statistical Analysis 1: Comparison: Study Group vs Control Group; Test type: Non-Inferiority — We hypothesized that Elonva 150 mcg is non-inferior for COH in obese women; p = 0.9, Regression, Logistic

2. Primary Outcome: Number of Mature Oocytes
Description: Number of mature oocytes obtained was compared between groups
Time Frame: 1 month
Measure: Number; unit: Mature oocytes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 35 | 35
Mature oocytes | 269 | 319
Statistical Analysis 1: Comparison: Study Group vs Control Group; Test type: Non-Inferiority — We hypothesized that Elonva 150 mcg is non-inferior for COH in obese women; p = 0.5, Regression, Logistic

3. Primary Outcome: Number of Fertilized Oocytes
Time Frame: 1 month
Measure: Number; unit: Fertilized oocytes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 35 | 35
Fertilized oocytes | 206 | 207
Statistical Analysis 1: Comparison: Study Group vs Control Group; Test type: Non-Inferiority — We hypothesized that Elonva 150 mcg is non-inferior for COH in obese women; p = 0.3, Regression, Logistic

4. Primary Outcome: Number of Frozen Embryos
Time Frame: 1 month
Measure: Number; unit: Frozen embryos
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 35 | 35
Frozen embryos | 45 | 49
Statistical Analysis 1: Comparison: Study Group vs Control Group; Test type: Non-Inferiority — We hypothesized that Elonva 150 mcg is non-inferior for COH in obese women; p = 0.9, Regression, Logistic

5. Primary Outcome: Biochemical Pregnancy Rate
Time Frame: 1 year
Measure: Number; unit: Biochemical pregnancies
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 35 | 35
Biochemical pregnancies | 18 | 18
Statistical Analysis 1: Comparison: Study Group vs Control Group; Test type: Non-Inferiority — We presumed Elonva 150 mcg in obese and normal weighing women yields comparable biochemical pregnancy rates; p = 0.4, Regression, Logistic

6. Secondary Outcome: Real-time PCR Analysis of Genes That Were Proposed as Biomarkers of Oocyte Quality to Determine Effect of Corifollitropin Alpha on Oocyte Quality on Molecular Level
Description: Expression of some genes that were proposed as biomarkers of oocyte quality was analysed in CC using real-time PCR. Relative expression values of genes were compared between mature oocytes derived from obese women and mature oocytes derived from normal weighing women.
Time Frame: 12 months
Population: Gene expression in cumulus cells surrounding mature oocytes was analyzed using quantitative polymerase chain reaction (qPCR). We analyzed 53 CC samples in the Study group and 56 CC samples in Control group.
Measure: Mean (Standard Deviation); unit: Arbitrary units (Relative expression)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 53 | 56
Arbitrary units (Relative expression)
  Progesterone receptor (PGR) | 2.52 (1.73) | 1.31 (0.9)
  Pentraxin 3 (PTX3) | 1.49 (1.37) | 0.63 (0.58)
  Serpin Family E Member 2 (SERPINE2) | 0.83 (0.75) | 0.61 (0.43)
  Follicle stimulating hormone receptor (FSHR) | 1.29 (1.58) | 1.2 (1.15)
  Glutathione peroxidase (GPX3) | 0.66 (1.31) | 0.33 (0.25)
  Hyaluronan Synthase 2 (HAS2) | 1.02 (0.78) | 0.96 (0.71)
  Versican (VCAN) | 5.40 (4.66) | 5.09 (5.6)
  Vascular endothelial growth factor C (VEGFC) | 0.79 (0.46) | 0.84 (0.42)

ADVERSE EVENTS:
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No